CLINICAL TRIAL: NCT03055923
Title: A Cross-sectional, Feasibility Study to Explore the Use of a New Device (Inflammacheck™) in Measuring the Level of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) in Patients With Asthma, COPD, and Healthy Volunteers. The EXHALE Pilot
Brief Title: EXhaled Hydrogen Peroxide As a Marker of Lung diseasE (EXHALE) Pilot Study.
Acronym: EXHALE Pilot
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Asthma UK (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2016/93
Record Dates: First submitted 2016-12-05; First posted 2017-02-16 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asthma Patients: 30 people who suffer from a confirmed diagnosis of asthma
  Interventions: Device: The Inflammacheck Device
- Chronic Obstructive Pulmonary Disease Patients: 30 people who suffer from a confirmed diagnosis of COPD
  Interventions: Device: The Inflammacheck Device
- Healthy Controls: 30 healthy volunteers who have no known diagnosis of Lung disease
  Interventions: Device: The Inflammacheck Device

INTERVENTIONS:
Device: The Inflammacheck Device — A new hand-held, Non-invasive breathing test, that only requires tidal breathing.

SUMMARY:
This Pilot study evaluates the use of a new device called Inflammacheck and whether it can consistently measure hydrogen peroxide levels in exhaled breath condensate. It will also assess whether exhaled breath condensate hydrogen peroxide levels as measured by Inflammacheck can differentiate people with asthma and COPD from healthy individuals.

DETAILED DESCRIPTION:
Hydrogen Peroxide levels in Exhaled Breath Condensate (EBC) is a direct biomarker of oxidative stress from the airway epithelium. Levels have been shown to be raised in asthma and Chronic Obstructive Pulmonary Disease (COPD) both in stable and exacerbating states.

Previously it has been difficult to measure this volatile compound away from a laboratory based setting. However a new device has been developed to measure Hydrogen peroxide levels in exhaled breath by the patients side.

This Pilot study will test this new device in a clinical setting. It will assess whether the device can monitor levels consistently and reliably and whether it can distinguish disease from healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinician made diagnosis of asthma with symptoms for ≥ 3 months supported by objective evidence of airflow variability, reversibility or airway hyper-responsiveness
* Subject has a confirmed, clinician made diagnosis of COPD for ≥ 3 months supported by spirometric evidence of fixed airflow limitation (post-bronchodilator ratio of FEV1/FVC <0.7) recorded at any time
* Subject has no known history of lung disease (defined as no current clinical diagnosis of, or be receiving treatment for, a lung disease).
* Subject is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Subject has existing co-morbidities that may prevent them from performing spirometry, FeNO or other study measurements (at the discretion of the clinical investigator).
* Subject has known other lung, chest wall, neuromuscular, or cardiac disease or abnormality (including end-stage disease or cancer) that would confound symptom scores and spirometry.
* Subject has received treatment for an exacerbation of their respiratory disease within the last 2 weeks.
* In the opinion of the clinical investigator, participant could be put at risk of harm by having to perform any of the study procedures.
* Subject is unable to comprehend the study and provide informed consent, e.g. insufficient command of English in the absence of someone to adequately interpret.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three populations of older adolescent and adult patients (all aged ≥16yrs) will be invited to participate:
  1. Asthma patients (n=30)
  2. COPD patients (n=30)
  3. Comparator group (n=30) - Volunteers with no previous history of lung disease.
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Exhaled Breath Condensate hydrogen peroxide levels as measured by the inflammacheck device. | 12 months

SECONDARY OUTCOMES:
Disease severity as measured by Global Initiative for Asthma (GINA) Stage for asthma. | 12 months
Disease severity as measured by Global Obstructive Lung Disease (GOLD) Stage for COPD. | 12 months
Disease control as measured by the Asthma Control Questionnaire (ACQ) score for asthma patients. | 12 months
Disease control as measured by the COPD Assessment Test (CAT) score for COPD patients. | 12 months
Quality of life as measured by the Asthma Quality of Life Questionnaire (AQLQ) score in asthma patients | 12 months
Lung function as recorded by the forced expiratory volume in 1 second (FEV1) | 12 months
Eosinophilic Lung Inflammation as recorded by the exhaled Nitric Oxide level (FeNO). | 12 months
Usability of inflammacheck device as measured by how frequently patients are unable to perform EBC collection by using the 'Inflammacheck' device. | 6 months
Acceptability of the inflammacheck device as measured by a questionnaire of the participants and healthcare professionals experience of 'Inflammacheck'. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Anoop J Chauhan, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, United Kingdom